CLINICAL TRIAL: NCT06682936
Title: Can Talc Pleurodesis for Malignant Pleural Effusion be Performed on an Ambulatory Basis
Brief Title: Feasibility of Ambulatory Talc. Pleurodesis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: David Rollins (Other)
Responsible Party: Sponsor-Investigator, David Rollins, Research governance manager - TVRA, North Tees and Hartlepool NHS Foundation Trust
Organization: North Tees and Hartlepool NHS Foundation Trust (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRAS:330188
Record Dates: First submitted 2024-01-10; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Malignant Pleural Effusion; Malignancy; Palliative Care
Keywords: malignant pleural effusion; malignancy; palliative care
MeSH Terms: conditions — Pleural Effusion, Malignant; Neoplasms

STUDY DESIGN:
Intervention Model Description: Feasibility of outpatient intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- outpatient drain and talc pleurodesis (Experimental): Patients enrolled to the trial will have a chest drain inserted and we will aim to drain to dryness and instill medical grade talc as described in the protocol
  Interventions: Procedure: ambulatory chest drain and talc pleurodesis

INTERVENTIONS:
Procedure: ambulatory chest drain and talc pleurodesis — a chest drain will be inserted, fluid drained and medical talc instilled on an ambulatory basis

SUMMARY:
Patients with malignant pleural disease often experience a significant symptom burden and a short life expectancy. The cornerstone of their treatment is relieving breathlessness by draining fluid from around the lungs and attempting to prevent further fluid build up. Inpatient chest drainage and talc pleurodesis remains the most successful method of stopping the fluid build up but this often requires an average hospital stay of four days. This can be an inappropriate length of time for this patient group. Our study would investigate whether this treatment could be provided on an outpatient, ambulatory basis and facilitate a greater quality of life.

The investigators would assess deliverability of the trial protocol and collect patient feedback to see if our patients consider it an acceptable and worthwhile intervention.

DETAILED DESCRIPTION:
Eligible patients will be offered enrolment in the trial along with standard of care options.

Participants who agree to take part in the trial would be consented for chest drain, talc pleurodesis on an ambulatory pathway.

On day 1 a standard chest drain would be inserted in the morning and large volume fluid removal would commence using an underwater seal bottle- as per standard care. A chest x-ray would be undertaken to confirm drain position, as per standard care. The investigators would remove 1000mls of fluid (stopping earlier if not tolerated) and the clamp the drain for one hour. The investigators would then open the drain again and drain up to 500mls before again clamping for one hour. The investigators would repeat this process as frequently as possible until the end of the working day. The drain would then be connected to an ambulatory bag instead of the underwater seal bottle and left in the open position. The patient would then be sent home to return on day 2.

On day 2 the drain would be flushed, aspirated and the output assessed. If there is still fluid output the investigators would drain up to 500mls and close the drain for an hour and repeat. If there is no further output the investigators would undertake a chest x ray to ensure the effusion has resolved and the lung has fully inflated. If it has the investigators would proceed to talc slurry instillation (with 20mls 1% lidocaine as per standard practice) and clamp the drain for 2 hours. After this the investigators would open the drain again and drain up to 500mls and close the drain for an hour. The investigators would repeat this as required and again the patient would return home with an ambulatory bag left open.

If the effusion has resolved but the lung has not fully expanded due to underlying disease then the investigators would simply remove the chest drain as pleurodesis will not be possible.

On day 3 the drain would be flushed, aspirated and the output assessed. If there is still fluid output the investigators would drain up to 500mls and close the drain for an hour and repeat. If there is no further output the investigators would undertake a chest x ray to ensure the effusion has resolved and the lung has fully inflated. the investigators would then remove the drain and repeat the x-ray to confirm there have been no complications. the investigators would then consider the intervention complete and revert to standard care (open access follow up )

If there was still significant fluid output the investigators would repeatedly drain 500ml volumes of fluid and clamp the drain for an hour after each 500ml until dry.

The investigators would ask patients to complete a very brief questionnaire (visual analogue scale) on breathlessness and chest pain on day 1 - before intervention, 1 hour post drain insertion, at the end of the day and on day 2 and 3 on first encounter and at the end of the day. The investigators would also repeat the questionnaire on day 30 along with their satisfaction with the procedure and if participants would have preferred to have stayed in hospital for the procedure (and why)

ELIGIBILITY:
Inclusion Criteria:

* Malignant pleural effusion
* Life expectancy >30 days
* WHO PS 1-2 (3 if due to dyspnoea)

Exclusion Criteria:

* Previous failed pleurodesis (on affected side)
* Known non-expansile lung

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-01-10 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Success rate of delivery of the ambulatory pleruodesis protocol | 5 days
  Can the investigators successfully deliver the described ambulatory pleruodesis protocol within the 5 day time frame and what is the success rate of the protocol delivery.

SECONDARY OUTCOMES:
Patient satisfaction / Patient related outcome measurement | 5 days
  Questionnaire on breathlessness and chest pain at day 5 and semi-structured interview on the patient experience of the intervention
Patient satisfaction / Patient related outcome measurement | 30 days
  Questionnaire on breathlessness and chest pain at day 30 and semi-structured interview of the patient experience of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Conroy, MBBS, FRCP, Principal Investigator — University Hospital of North Tees
Locations (1):
- North Tees and Hartlepool NHS foundation trust, Stockton-on-Tees, County Durham, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The primary end point of this trial is feasibility of intervention delivery. We will share our results and our protocol. All other outcomes are qualitative and will be reported at the end of the trial. Making individual participant data available to other researches does not seem necessary

DOCUMENTS (1):
  • Study Protocol (2023-06-26): https://cdn.clinicaltrials.gov/large-docs/36/NCT06682936/Prot_000.pdf